CLINICAL TRIAL: NCT02639806
Title: General Anesthesia for Endovascular Thrombectomy; A Pilot Study.
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Michael Kelly, Professor, MD, PHD, University of Saskatchewan
Other Study IDs: SEVO-01
Record Dates: First submitted 2015-12-18; First posted 2015-12-24 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Stroke; Cerebrovascular Stroke; Brain Ischemia; Brain Diseases; Cardiovascular Diseases; Central Nervous System Diseases; Cerebrovascular Disorders; Nervous System Diseases; Vascular Diseases
Keywords: stroke; endovascular; thrombectomy; ischemic stroke; general anesthetic; local anesthetic; recanalization
MeSH Terms: conditions — Stroke; Brain Ischemia; Brain Diseases; Cardiovascular Diseases; Central Nervous System Diseases; Cerebrovascular Disorders; Nervous System Diseases; Vascular Diseases; Ischemic Stroke | interventions — Sevoflurane; Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective - General Anesthetic: The prospective treatment group will have an anesthetic induction according to the anesthetic provider's preference that will include propofol and fentanyl as IV induction agents and rocuronium as a muscle paralytic. Maintenance of anesthesia for the treatment group will include sevoflurane with a target end tidal concentration of 1-1.5%, rocuronium as a paralytic as needed, opioids and any other standard medication deemed necessary by the provider.
  Interventions: Drug: Sevoflurane
- Retrospective - Local Anesthetic with Sedation: The retrospective group will have received local anesthetic from the surgeon using lidocaine injected subcutaneously and received sedation using fentanyl and midazolam as needed to achieve the desired level of sedation.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Sevoflurane
  Groups: Prospective - General Anesthetic
Drug: Lidocaine
  Groups: Retrospective - Local Anesthetic with Sedation

SUMMARY:
This study evaluates the outcomes of stroke patients treated for intravascular thrombectomy, using either a local anesthetic with sedation, or a general anesthetic. Historical data will be used for those treated with the local anesthetic, and prospective data will be used for those treated with the general anesthetic.

DETAILED DESCRIPTION:
This is an open-label pilot study, comparing intravascular thrombectomy patients treated using either general anesthetic (prospective arm) or local anesthetic with sedation (retrospective arm), with blinded outcome evaluation.

New evidence has established that the addition of endovascular thrombectomy for large, and/or proximal occlusions improves outcome in addition to, and/or in place of tPA therapy. There have been no randomized prospective trials assessing the relationship of anesthesia on outcomes for this procedure. This procedure is routinely performed under either local anesthetic with sedation and under general anesthesia (GA). The choice between these two techniques is largely institution based. Currently in the Saskatoon Health Region (SHR) endovascular thrombectomies are performed under general anesthesia due to operator preference and the optimization of surgical conditions. In the United States and other Canadian centers, this procedure is performed safely with local anesthesia with or without sedation.

Several retrospective trials have suggested that general anesthetics are associated with poorer outcomes. It has been suggested that general anesthesia can result in a delay in the time to procedural start since it requires the presence of an anesthesiologist and the procedure can be performed under sedation without extra personnel. It is also proposed that the induction of general anesthesia can cause a decrease in blood pressure and a decrease in collateral perfusion which can result in further cellular hypoxia. Anesthesiologists , however, are able to expertly manipulate hemodynamic parameters during general anesthesia to the specific requirements of the operators potentially creating optimal tissue oxygenation conditions.

There is a need for a prospective trial to assess the effect of general anesthetic on patient outcome during endovascular thrombectomy. At this time, it is premature to conduct a randomized controlled trial (RCT). Therefore in this pilot study, adult acute ischemic stroke participants who undergo intravascular thrombectomy in Saskatchewan will receive a general anesthetic as per their current practice, and their data will be collected prospectively. This cohort of participants will then be compared to participants that underwent the same procedure in another study, who received local anesthesia with sedation. Approximately 77 prospective participants will be recruited for the prospective arm of this study.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Age 18 or greater
* Onset (last seen well) time to treatment less than 12 hours
* Disabling stroke defined as a baseline NIHSS > 5 at the time of treatment
* Pre-stroke independent functional status in activities of daily living. Patient must be living in their own home, apartment or seniors lodge where no nursing care is required
* Pre-enrollment non-intubated state based on acceptable GCS for the prospective Cohort
* Small core proximal occlusion as confirmed by CT angiography (carotid, M1 MCA or M1 MCA equivalent)
* Intention to initiate endovascular treatment within 60 minutes of baseline non-contrast CT
* Sevoflurane used during thrombectomy
* Appropriate consent provided

Exclusion Criteria:

* Baseline non-contrast CT reveals a moderate/large core defined as extensive early ischemic changes of ASPECTS 0-5 in the territory of symptomatic intracranial occlusion
* Hemorrhagic stroke
* Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic
* Intubated state based on GCS at any time prior to induction of general anesthesia for prospective cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult acute ischemic stroke participants who undergo intravascular thrombectomy in Saskatchewan will be prospectively recruited for the prospective arm.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Shift in the mRS score, defined by a proportional odds model. | 90 Days

SECONDARY OUTCOMES:
The proportion of patients who achieve a NIHSS score 0-2 | 90 Days
  Stroke severity. Clinical scale outcome score from 0 to 42.
The proportion of patients who achieve a mRS 0-2 | 90 days
  Functional outcome. Dichotomous outcome, reported as independent (mRS 0-2) vs dependence or death (mRS 3-6). In addition, shift analysis (proportional odds model) representing the odds of improvement within the scale with treatment.
Recanalization of the target arterial occlusive lesion | Day 0
  Measured by fluoroscopy - Demonstrated during (or as part of) the procedure.
Time from diagnostic CT to procedure initiation | Day 0
Time from the start of the procedure to vascular recanalization | Day 0
Incidence of Treatment-Emergent Adverse Events | 90 Days
  Episodes of hypo/hypertensive and bradycardic episodes that required the use of pharmacologic agent.; Symptomatic intracranial hemorrhage; Major bleeding; Contrast nephropathy; Malignant MCA infarction; Hemicraniectomy; Aspiration Pneumonia; Adverse airway event; other

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kelly, MD, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada